CLINICAL TRIAL: NCT00960466
Title: Evaluating the Effect of Monitoring Cancer Patients Using the Distress Thermometer on Levels of Distress and Health Service Costs - a Randomised Controlled Trial
Brief Title: Distress Thermometer Intervention Trial
Acronym: DiTIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: Royal United Hospital Bath NHS Trust (Other); University of Bristol (Other)
Responsible Party: Principal Investigator, William Hollingworth, Reader, School of Social and Community Medicine, University Hospitals Bristol and Weston NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ON/2007/2744; REC # 08/H0101/224; NIHR # PB-PG-0807-13387
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Cancer
Keywords: Stress, Psychological; Neoplasms/psychology; Psychology
MeSH Terms: conditions — Neoplasms; Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Arm (Active Comparator): The usual care group will receive their Chemotherapy or Radiotherapy as normal.
  Interventions: Behavioral: Usual psychosocial support
- DT&PL arm (Experimental): During the second week of radiotherapy/second cycle of chemotherapy, patients in the Distress Thermometer and Problem List (DT&PL) arm of the study will complete the DT&PL (estimated 15 minutes to complete) with the trained radiographer/nurse.
  The DT&PL assessment will be repeated at the end of therapy fractions/cycles. This will elicit concerns about post-therapy issues and facilitate continuity of care between the cancer team and primary care. Depending on the duration of therapy, therapists may choose to use the DT&PL at other points during patient care. A copy of the DT&PL will be stored in the medical record to track the frequency of use and to check that those assigned to usual care were not monitored with the DT&PL.
  Interventions: Behavioral: Distress Thermometer and Problems List

INTERVENTIONS:
Behavioral: Distress Thermometer and Problems List — When using the distress thermometer and problem list (DT&PL), the nurse or radiographer asks the patient to indicate distress over the past week on a visual analogue scale from 0 (no distress) to 10 (high distress). Next, from a list of 42 items, patients identify practical, family, emotional, spiritual or physical problems that have caused distress. The completion of the DT&PL should be a collaborative exercise with patients able to review what is written on the assessment sheet. Potential solutions will be discussed which may involve the following: i) concerns that can be resolved immediately (e.g. providing information, prescribing an analgesic); ii) concerns that require patient actions (e.g. participating in support groups); iii) concerns that require a referral (e.g. mental health specialist, social or pastoral care). The meeting will end with a summary plan of action.
  Arms: DT&PL arm
Behavioral: Usual psychosocial support — If patients express concerns about psychosocial issues, then clinic staff will discuss these issues, offer advice or make a referral as they see fit. However, no formal time will be set aside to monitor patient distress using the DT, elicit problems using the PL or develop a plan of action based on these tools. Because of the nature of the intervention, both the patient and the therapist will be aware of treatment assignment.
  Arms: Usual Care Arm

SUMMARY:
The diagnosis and treatment of cancer has been shown to lead to very high levels of distress among patients. Although treatments for a range of different cancers have become much better in recent years, the distress that accompanies diagnosis and treatment can have serious negative effects for patients. Research has shown that, for a number of reasons, patients find it difficult to inform healthcare professionals about the cause of their distress whether it is physical (e.g. pain), psychological (anxiety and depression), personal partners and family) or social (finances). Also, medical staff often fail to detect even high levels of distress. This means that a great deal of distress is not being treated and this may lead to more hospital and GP visits, and dissatisfaction with care. The Distress Thermometer and Problem List (DT&PL) is a simple method of identifying distress in cancer patients using the familiar image of a thermometer. It offers patients a list of common treatment-related difficulties to help them identify any problems that cause distress. A trained staff member uses the DT&PL to discuss with the patient different options for addressing each concern: directly where possible (action taken by the patient or the staff member present) or leading to a referral to a specialist where necessary. Our research aims to measure whether the DT&PL is effective in quickly identifying and treating cancer-related distress and therefore preventing longer-term problems developing. The investigators also want to know whether patients find it helpful to complete the DT&PL and whether using the DT&PL saves NHS time and money.

DETAILED DESCRIPTION:
BACKGROUND: Systematic psychological assessment and appropriate psychological support is a key aim of NICE guidance for supportive and palliative cancer care. Cancer causes high levels of distress during diagnosis, treatment and beyond. 'Distress' is a psychological state that may be fuelled by physical (e.g. pain), interpersonal (family tensions), psychological (anxiety and depression), social (finances), and existential concerns. Often these concerns are not expressed by patients or identified by healthcare staff. Our pilot work suggests that the Distress Thermometer and Problem List (DT&PL) is a tool that healthcare staff can use to efficiently identify and address these holistic needs. Use of the DT&PL could reduce both patient distress and the NHS costs of treating the sequelae of distress.

AIMS: To demonstrate the feasibility of performing a randomised controlled trial (RCT) in 3 cancer therapy units and to provide data for the design of a future trial in larger numbers of radiotherapy and chemotherapy units. To compare use of the Distress Thermometer and Problem List (DT&PL) with usual care and document differences in patients' psychological well-being and health-related quality of life. To assess the cost-effectiveness to the NHS and society of using the DT&PL in routine clinical practice. To assess patient and staff attitudes to completing the DT&PL and identify any perceived gaps in local psychosocial supportive services.

METHODS: A RCT to compare usual psychosocial care with usual care plus DT&PL administered by trained radiographers and nurses for cancer patients receiving chemotherapy or radiotherapy. The DT&PL will be used during and at the end of chemo/radiotherapy. Baseline questionnaires include Profile of Mood States (POMS - primary outcome), European Organisation for Research and Treatment of Cancer (EORTC) cancer-related quality of life measure and EQ-5D utility score. Qualitative interviews will explore patient, carer and staff views on the DT&PL and other aspects of supportive care. Patient follow up will occur at 1, 6 and 12 months to determine whether the intervention improves psychological well-being and health related quality of life and the impact on NHS and broader societal costs.

ELIGIBILITY:
Inclusion Criteria:

* Primary solid tumour diagnosis within the last 12 months
* Scheduled for outpatient external RT fractions over a period of at least 2 weeks or scheduled outpatient CT regimen over 2 or more cycles
* Patient aged >= 18 and <85 years
* Ability to read and communicate in English (personally or via translator)

Exclusion Criteria:

* Receiving neoadjuvant CT
* Patient declines consent
* Clinical presentation dictates treatment by a specific therapist not trained in use of the Distress Thermometer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States (POMS) | 1, 6, 12 months post randomisation

SECONDARY OUTCOMES:
EQ-5D | 1,6,12 months post randomisation
European Organisation for Research and Treatment of Cancer (EORTC - QLQ 30) cancer-related quality of life measure | 1,6, 12 months post randomisation
Trent Patient Satisfaction Questionnaire | 1, 6 months post randomisation
Resource Use | 12 months post randomisation
Mortality | 12 months post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: William Hollingworth, PhD, Principal Investigator — University of Bristol
Locations (2):
- United Kingdom (2):
  - Royal United Hospital, Bath, Somerset
  - University Hospitals Bristol, Bristol

REFERENCES:
- [Background] Brennan J, Gingell P, Brant H, Hollingworth W. Refinement of the distress management problem list as the basis for a holistic therapeutic conversation among UK patients with cancer. Psychooncology. 2012 Dec;21(12):1346-56. doi: 10.1002/pon.2045. Epub 2011 Sep 9. PMID 21905157
- [Result] Hollingworth W, Metcalfe C, Mancero S, Harris S, Campbell R, Biddle L, McKell-Redwood D, Brennan J. Are needs assessments cost effective in reducing distress among patients with cancer? A randomized controlled trial using the Distress Thermometer and Problem List. J Clin Oncol. 2013 Oct 10;31(29):3631-8. doi: 10.1200/JCO.2012.48.3040. Epub 2013 Sep 3. PMID 24002506